CLINICAL TRIAL: NCT02403323
Title: An Open-Label Extension and Safety Monitoring Study of Patients With Moderately to Severely Active Crohn's Disease Previously Enrolled in the Etrolizumab Phase III Protocol GA29144
Brief Title: Open-Label Extension and Safety Study for Participants With Crohn's Disease Previously Enrolled in the Etrolizumab Phase III Study GA29144
Acronym: JUNIPER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to program discontinuation, based on mixed efficacy results in the parent studies. There were no safety concerns.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA29145; 2014-003855-76 (EudraCT Number)
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — etrolizumab

ARMS (2):
- Part 1: Etrolizumab Open-Label Extension (Experimental): Participants will receive open-label treatment with etrolizumab once every 4 weeks until commercial availability in their country or sponsor's decision to terminate the study, whichever is earlier (up to approximately 10 years after the first patient is enrolled).
  Interventions: Drug: Etrolizumab
- Part 2: Safety Monitoring (No Intervention): Participants who have stopped etrolizumab treatment (either by exiting Part 1 of this study or by entering directly from Study GA29144 [NCT02394028]) will be monitored for 92 weeks for progressive multifocal leukoencephalopathy (PML) and other safety events.

INTERVENTIONS:
Drug: Etrolizumab — 105 mg etrolizumab subcutaneous administration once every 4 weeks
  Other Names: RG7413
  Arms: Part 1: Etrolizumab Open-Label Extension

SUMMARY:
This open-label extension and safety monitoring study is composed of two parts: Part 1 will evaluate the long-term safety and efficacy of continued etrolizumab treatment in participants with moderately to severely active Crohn's disease who were previously enrolled in the etrolizumab Phase III Study GA29144 (NCT02394028) and who meet eligibility criteria for enrollment into Part 1. In Part 2, participants who have stopped etrolizumab treatment (either by exiting Part 1 of this study or by entering directly from Study GA29144 [NCT02394028]) will be monitored for 92 weeks for progressive multifocal leukoencephalopathy (PML) and other safety events.

ELIGIBILITY:
Inclusion Criteria:

Part 1 Open-Label Extension:

* Patients previously enrolled in etrolizumab Phase III study GA29144 (NCT02394028) who meet the eligibility criteria for open-label etrolizumab as described in the protocol

Part 2 Safety Monitoring:

* Patients who participated in etrolizumab Phase III study GA29144 (NCT02394028) and are not eligible or choose not to enter Part 1
* Patients who transfer from Part 1
* Completion of the 12-week safety follow-up period prior to entering

Exclusion Criteria:

Part 1 Open-Label Extension:

* Any new, significant, uncontrolled condition

Part 2 Safety Monitoring:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (287):
- United States (59):
  - Valley Gastroenterology Consultants, Arcadia, California
  - University of California San Diego Medical Center, La Jolla, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Digestive Care Associates, A Medical Corporation, San Carlos, California
  - SDG Clinical Research, San Diego, California
  - Uni. of California at San Francisco; Dept Pediatric, Div. of Gastroenterology, Hepatology & Nutri, San Francisco, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Innovative Medical Research of South Florida, Aventura, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - IMIC, Inc, Miami Beach, Florida
  - FQL Research, LLC, Miramar, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Atlanta Center for Gastroenterology, PC, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Advanced Clinical Research, Spokane, Idaho
  - Northwestern Uni-Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Grand Rapids, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Concorde Medical Group, New York, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Vidant Medical Group, LLC DBA Vidant Multispeciality Clinic-Kinston, Kinston, North Carolina
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Great Lakes Medical Research, LLC, Harrisburg, Pennsylvania
  - Innovative Clinical Research, Greenville, South Carolina
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center; Internal Medicne, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Methodist Hospital Research Institute, Houston, Texas
  - Wellness Clinical Research Center, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Ericksen Research and Development, Clinton, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - McGuire Research Institute; Gastroenterology, Richmond, Virginia
  - Digestive Disease Institute; Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Hospital Italiano, CABA, Argentina
- Australia (13):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - St Frances Xavier Cabrini Hospital, Malvern, Victoria
  - Royal Melbourne Hospital; Department of Colorectal Medicine and Genetics, Parkville, Victoria
  - The Alfred Hospital, Prahan, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (2):
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (5):
  - CHU St Pierre (César de Paepe) X, Brussels
  - ULB Hopital Erasme; Service de Néphrologie, Brussels
  - UZ Brussel, Brussels
  - UZ Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
- Brazil (15):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Instituto Brasil de Pesquisa Clínica-IBPCLIN S/A, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Pesquisare Saúde Sociedade Simples, Santo André, São Paulo
  - Praxis Pesquisa Médica, Santo André, São Paulo
  - Hospital Estadual Mario Covas, São Bernardo do Campo, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFES, São Paulo, São Paulo
  - Hospital do Servidor Público Estadual/HSPE-SP, São Paulo, São Paulo
- Bulgaria (2):
  - "City Clinic UMHAC" EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
- Canada (13):
  - University of Calgary, Calgary, Alberta
  - Zeidler Ledcor Centre - University of Alberta; Division of Gasroenterology, Edmonton, Alberta
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Winnipeg Regional Health Authority; Neurosurgery Department, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre; Gastroenterology Research, Halifax, Nova Scotia
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Taunton Health Centre, Oshawa, Ontario
  - The Ottawa Hospital - Riverside Campus; Gastrointestinal Clinical Research Unit, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Croatia (3):
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Pula, Pula
  - Clinical Hospital Center Sestre Milosrdnice, Zagreb
- Czechia (10):
  - Vojenska nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne; I.Interni kardioangiologicka klinika, Brno
  - Nemocnice Ceske Budejovice a.s., České Budějovice
  - Gastroenterologie s.r.o., Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - PreventaMed, s.r.o., Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - ISCARE a.s., Prague
- Estonia (3):
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- France (13):
  - CHU Amiens - Hopital Sud, Amiens
  - CHU de Caen Hopital Cote de Nacre, Caen
  - Hôpital Beaujon, Clichy
  - Hopital Claude Huriez - CHU Lille, Lille
  - CHU NANTES - Hôtel Dieu; Pharmacy, Nantes
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Hôpital Saint-Louis, Paris
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - USN, Pessac
  - Centre Hospitalier Lyon Sud; Service de Gastro-Enterologie, Pierre-Bénite
  - CHU du Reims - Hopital Robert Debré, Reims
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Höpital Hautepierre; Pediatrie1, Strasbourg
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (8):
  - Charite-Campus Virchow Klinikum; Hepatologie und Gastroenterologie, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
  - Berufsgenossenschaftliches Universitaetsklinikum Bergmannsheil GmbH, Bochum
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Gemeinschaftspraxis, Schweinfurt
  - Universitaetsklinikum Ulm, Ulm
- Hungary (8):
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaza, Békéscsaba
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem; Belgyogyaszati es Hematologiai Klinika, Budapest
  - Szt Janos Korhaz es EbudaiEgyesitettKorhazak, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Debreceni Egyetem Klinikai Központ; B?rgyógyászati Klinika, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
- Israel (7):
  - Haemek Medical Center, Afula
  - Soroka University Medical Centre, Beersheba
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center; Pharmacy, Tel Aviv
- Italy (7):
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Policlinico Universitario Agostino Gemelli; Farmacia, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Asst Fatebenefratelli Sacco (Fatebenefratelli), Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese (MI), Lombardy
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, R?ga
  - Riga East Clinical University Hospital, clinic "Gailezers"; Department of Endoscopy, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santariskiu Clinics, Public Inst; Department of Clinical Pharmacology, Vilnius
- Mexico (2):
  - Clinical Research Institute, Tlalnepantla, Mexico CITY (federal District)
  - Medical Care & Research SA de CV, Mérida, Yucatán
- Netherlands (7):
  - Amsterdam UMC, Locatie VUMC; Gastroenterology, Amsterdam
  - Amsterdam UMC Location AMC, Amsterdam
  - Leids Universitair Medisch Centrum; Cardiology, Leiden
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
  - ETZ TweeSteden, Tilburg
- New Zealand (7):
  - North Shore Hospital, Auckland
  - Christchurch Hospital NZ, Christchurch
  - Dunedin Public Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Hutt Hospital, Lower Hutt
  - Shakespeare Specialist Group, Takapuna
  - Tauranga Hospital, Tauranga
- Poland (17):
  - SP ZOZ Wojewodzki Szpital Zespolony im. J. Sniadeckiego, Bia?ystok
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Elblaski Szpital Specjalistyczny z Przychodnia SP ZOZ, Elblag
  - ETG Kielce, Kielce
  - Centrum Opieki Zdrowotnej Orkan-Med, Ksawerów
  - Indywidualna Specjalistyczna Praktyka Lekarska, Lublin
  - Allmedica Badania Kliniczne Sp z o.o. Sp K., Nowy Targ
  - Centrum Medyczne "MEDYK", Rzeszów
  - Gabinet Lekarski, Bartosz Korczowski, Rzeszów
  - Niepubliczny Zaklad Opieki Zdrowotnej SONOMED, Szczecin
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Gastromed Kopon Zmudzinski i Wspolnicy Sp.j.Specjalistyczne Centrum Gastrologii i Endoskopii Specj, Toru?
  - Centrum Zdrowia MDM, Warsaw
  - Zespó Przychodni Specjalistycznych PRIMA, Warsaw
  - Przychodnia EuroMediCare, Wroc?aw
  - PlanetMed sp. z o.o., Wroc?aw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
- Romania (3):
  - S.C MedLife S.A, Bucharest
  - Spitalul Clinic Colentina, Sector 2
  - Centrul de Gastroenterologie Dr. Goldis, Timișoara
- Russia (12):
  - LLC "Novosibirsk GastroCenter", Novosibirsk, Altaj
  - SBEI HPE Altai StateMedicalUniversityofMoH andSD, Barnaul, Altayskiy Kray
  - LEC at SBIH of Moscow "City Clinical Hospital # 24"; Gastroenterology, Moscow, Moscow Oblast
  - SEIHPE "Rostov SMU of MoH of RF", Rostov-on-Don, Rostov Oblast
  - Evromedservis LCC, Pushkin, Sankt-Peterburg
  - Federal State Military Educational Inst. of High Prof. Edu Military Medical Acad; Therapy department, Saint Petersburg, Sankt-Peterburg
  - North-Western Medical University n.a. I.I. Mechnikov; Rheumatology, Saint Petersburg, Sankt-Peterburg
  - Baltic Medicine, Saint Petersburg, Sankt-Peterburg
  - SBIH City Clinical Hospital #31, Saint Petersburg, Sankt-Peterburg
  - Irkutsk State Medical Academy of Continuing Education, Irkutsk
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
- Serbia (3):
  - Clinical Center Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - General Hospital Djordje Joanovic, Zrenjanin
- Slovakia (3):
  - Endomed, s.r.o., Košice
  - KM Management spol. s r.o., Nitra
  - Accout Center s.r.o., Šahy
- South Africa (2):
  - Dr D Epstein Practice, Cape Town
  - Emmed Research, Pretoria
- South Korea (10):
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam Univ. Hospital, Daegu
  - Korea University Ansan Hospital, Gyeonggi-do
  - CHA Bundang Medical Centre; CHA university, Seongnam
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (11):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic i Provincial; Servicio de Farmacia, Barcelona
  - Hospital Reina Sofia; Medical Oncology, Córdoba
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Inselspital-Universitaetsspital Bern, Bern
  - Crohn-Colitis Zentrum Bern - Gemeinschaftspraxis Balsiger, Seibold und Partner, Bern
  - Universitätsspital Zürich, Zurich
- Turkey (Türkiye) (7):
  - Hacettepe University Medical Faculty; Gastroenterology, Ankara
  - Gazi University Medical Faculty, Ankara
  - Acibadem Fulya Hospital; Neurology, Istanbul
  - Haydarpasa Numune Training and Research Hospital; Gastroenterology, Istanbul
  - Medeniyet University Goztepe Training and Research Hospital., Kadiköy
  - Kocaeli Universitesi Tip Fakultesi; Infectious Diseases, Kocaeli
  - Acibadem Kozyatagi Hospital; Gastroenterology, Kozyata?i
- Ukraine (14):
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv, Kharkiv Governorate
  - CI of Healthcare Kharkiv Reg Clin Hosp-Center of Med Emergency & Accident Medicine, Kharkiv, Kharkiv Governorate
  - LLC Gastroenterology Center IBD Team, Zaporizhzhia, Kharkiv Governorate
  - Medical Center of Limited Liability Company Medical Clinic Blagomed, Kyiv, KIEV Governorate
  - Med Center of International Institute of Clinical Trials LLC; Medical Center "OK!Clinic+", Kyiv, KIEV Governorate
  - CI of Kyiv RC Regional Clinical Hospital #2, Kyiv, KIEV Governorate
  - Lviv Regional Clinical Hospital, Lviv, KIEV Governorate
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk, Kuban People's Republica
  - RCI Chernivtsi RCH Dep of Surgery Bukovinian SMU, Chernivtsi
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - Railway Transport Odesa CH of Healthcare Ctr Branch of PJSC Ukrainian Railway Dept of Therapy #2, Odesa
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
- United Kingdom (13):
  - Royal Victoria Hospital, Belfast
  - University Hospital Coventry, Coventry
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Queen Elizabeth Hospital, Kings Lynn
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Whipps Cross Hospital, London
  - University College London Hospital, London
  - Fairfield General Hospital, Manchester
  - Royal Victoria Infirmary; Stroke unit, Newcastle upon Tyne
  - Nottingham University Hospitals Queen's Medical Centre, Nottingham
  - Royal Berkshire Hospital, Reading
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Sandborn WJ, Vermeire S, Tyrrell H, Hassanali A, Lacey S, Tole S, Tatro AR; Etrolizumab Global Steering Committee. Etrolizumab for the Treatment of Ulcerative Colitis and Crohn's Disease: An Overview of the Phase 3 Clinical Program. Adv Ther. 2020 Jul;37(7):3417-3431. doi: 10.1007/s12325-020-01366-2. Epub 2020 May 22. PMID 32445184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study in 33 countries. All participants who enrolled into this study previously took part in study GA29144 (NCT02394028).
Pre-assignment Details: This study consists of 2 parts, Part 1: Open-label extension (OLE) period & Part 2: Progressive multifocal leukoencephalopathy (PML) safety monitoring (SM) period. A total of 790 participants were enrolled in the study, 751 participants in Part 1 and 359 participants in Part 2. Of the 359, 39 participants directly entered into the Part 2 PML SM period from study GA29144.
Groups:
- Part 1 (OLE): Etrolizumab Only: Participants received etrolizumab 105 milligrams (mg), subcutaneously (SC), once every 4 weeks (Q4W) for a maximum of 320 weeks followed by a 12-week safety follow-up.
- Part 1 (OLE) to Part 2 (PML SM): Participants received etrolizumab 105 mg, SC, Q4W for maximum of 320 weeks, followed by a 12-week safety follow-up in the OLE period. After the OLE period, participants were given the option to enter Part 2 (PML SM). Participants who chose to enter the PML SM period were monitored for PML for a maximum of 92-weeks, during which no etrolizumab treatment was administered.
- Part 2 (PML SM) Only: Participants from study GA29144 who completed the 12-week safety follow-up period and were not eligible/did not wish to enroll in the Part 1 (OLE), enrolled directly in Part 2 (PML SM). Participant were monitored for PML for a maximum of 92-weeks, during which no etrolizumab treatment was administered.
Period: Part 1: Open Label Extension Period
Arm/Group | Part 1 (OLE): Etrolizumab Only | Part 1 (OLE) to Part 2 (PML SM) | Part 2 (PML SM) Only
Started | 431 | 320 | 0
Completed | 5 | 320 | 0
Not Completed | 426 | 0 | 0
Not completed — Adverse Event | 26 | 0 | 0
Not completed — Death | 3 | 0 | 0
Not completed — Lost to Follow-up | 23 | 0 | 0
Not completed — Non-Compliance | 2 | 0 | 0
Not completed — Reason Not Specified | 59 | 0 | 0
Not completed — Physician Decision | 61 | 0 | 0
Not completed — Study Terminated By Sponsor | 19 | 0 | 0
Not completed — Other | 1 | 0 | 0
Not completed — Withdrawal by Subject | 232 | 0 | 0
Period: Part 2: PML Safety Monitoring Period
Arm/Group | Part 1 (OLE): Etrolizumab Only | Part 1 (OLE) to Part 2 (PML SM) | Part 2 (PML SM) Only
Started | 0 | 320 | 39
Completed | 0 | 112 | 33
Not Completed | 0 | 208 | 6
Not completed — Adverse Event | 0 | 4 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 9 | 3
Not completed — Non-Compliance | 0 | 1 | 0
Not completed — Reason Not Specified | 0 | 6 | 1
Not completed — Physician Decision | 0 | 7 | 0
Not completed — Study Terminated By Sponsor | 0 | 167 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 12 | 2

BASELINE CHARACTERISTICS:
Population: All Patients Population included all participants who were enrolled in the study.
Groups:
- Part 1 (OLE): Etrolizumab Only: Participants received etrolizumab 105 mg, SC, Q4W for a maximum of 320 weeks followed by a 12-week safety follow-up.
- Total: Total of all reporting groups
Arm/Group | Part 1 (OLE): Etrolizumab Only | Part 1 (OLE) to Part 2 (PML SM) | Part 2 (PML SM) Only | Total
Number analyzed (Participants) | 431 | 320 | 39 | 790
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (13.0) | 39.7 (13.6) | 36.8 (13.0) | 38.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 158 | 19 | 376
  Male | 232 | 162 | 20 | 414
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 3 | 51
  Not Hispanic or Latino | 385 | 280 | 35 | 700
  Unknown or Not Reported | 22 | 16 | 1 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 0 | 4
  Asian | 25 | 8 | 2 | 35
  Black or African American | 15 | 10 | 2 | 27
  White | 358 | 277 | 33 | 668
  Multiple | 2 | 1 | 0 | 3
  Unknown | 21 | 14 | 1 | 36
  Other | 10 | 6 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Crohn's Disease Activity Index (CDAI) Remission at 12-week Intervals
Description: CDAI is a score obtained from composite of eight assessments: number of liquid or soft stools, abdominal pain, general well-being, presence of complications, taking lomotil (diphenoxylate/atropine) or other opiates for diarrhea, presence of an abdominal mass, hematocrit, and percentage deviation from standard weight. A decrease in CDAI over time indicates improvement in disease activity. CDAI scores range from 0 to 600. A higher score indicates worse outcome. A total score of less than 150 corresponds to remission.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240 and 252 of OLE
Population: OLE population included all participants who received at least one dose of study drug in Study GA29145 Part 1 (OLE). Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 (OLE): Etrolizumab: Participants received etrolizumab 105 mg, SC, Q4W for a maximum of 320 weeks followed by a 12-week safety follow-up.
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants
  Day 1 | 230
  Week 12: number analyzed (Participants) | 354
  Week 12 | 166
  Week 24: number analyzed (Participants) | 285
  Week 24 | 165
  Week 36: number analyzed (Participants) | 250
  Week 36 | 161
  Week 48: number analyzed (Participants) | 163
  Week 48 | 113
  Week 60: number analyzed (Participants) | 198
  Week 60 | 137
  Week 72: number analyzed (Participants) | 180
  Week 72 | 124
  Week 84: number analyzed (Participants) | 160
  Week 84 | 119
  Week 96: number analyzed (Participants) | 119
  Week 96 | 88
  Week 108: number analyzed (Participants) | 123
  Week 108 | 96
  Week 120: number analyzed (Participants) | 109
  Week 120 | 85
  Week 132: number analyzed (Participants) | 97
  Week 132 | 73
  Week 144: number analyzed (Participants) | 87
  Week 144 | 62
  Week 156: number analyzed (Participants) | 80
  Week 156 | 58
  Week 168: number analyzed (Participants) | 81
  Week 168 | 57
  Week 180: number analyzed (Participants) | 73
  Week 180 | 53
  Week 192: number analyzed (Participants) | 50
  Week 192 | 39
  Week 204: number analyzed (Participants) | 46
  Week 204 | 29
  Week 216: number analyzed (Participants) | 44
  Week 216 | 32
  Week 228: number analyzed (Participants) | 33
  Week 228 | 18
  Week 240: number analyzed (Participants) | 24
  Week 240 | 13
  Week 252: number analyzed (Participants) | 21
  Week 252 | 12

2. Primary Outcome: Part 1: Number of Participants With Clinical Remission at 12-week Intervals
Description: Clinical remission was defined as a liquid/soft stool frequency (SF) mean daily score ≤3 and an abdominal pain (AP) mean daily score ≤1 with no worsening in either subscore compared to baseline, where the average was taken over 7 days prior to visit. Abdominal pain severity was assessed using the abdominal pain questionnaire which is an 11-point numeric rating scale with score ranging from 0 (no pain) to 10 (worse pain). Liquid/soft stool frequency was reported using the bristol stool form scale which classifies stools into seven groups based on its consistency i.e., type 1- separate hard lumps, type 2- sausage-shaped but lumpy, type 3- like a sausage but with cracks on the surface, type 4- like a sausage or snake, smooth and soft, type 5- soft blobs with clear-cut edges, type 6- fluffy pieces with ragged edges and type 7- entirely liquid with no solid pieces.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants
  Day 1 | 200
  Week 12: number analyzed (Participants) | 397
  Week 12 | 161
  Week 24: number analyzed (Participants) | 346
  Week 24 | 168
  Week 36: number analyzed (Participants) | 302
  Week 36 | 162
  Week 48: number analyzed (Participants) | 244
  Week 48 | 135
  Week 60: number analyzed (Participants) | 231
  Week 60 | 131
  Week 72: number analyzed (Participants) | 221
  Week 72 | 132
  Week 84: number analyzed (Participants) | 193
  Week 84 | 119
  Week 96: number analyzed (Participants) | 171
  Week 96 | 103
  Week 108: number analyzed (Participants) | 141
  Week 108 | 89
  Week 120: number analyzed (Participants) | 128
  Week 120 | 87
  Week 132: number analyzed (Participants) | 116
  Week 132 | 71
  Week 144: number analyzed (Participants) | 106
  Week 144 | 71
  Week 156: number analyzed (Participants) | 102
  Week 156 | 64
  Week 168: number analyzed (Participants) | 97
  Week 168 | 62
  Week 180: number analyzed (Participants) | 88
  Week 180 | 57
  Week 192: number analyzed (Participants) | 67
  Week 192 | 41
  Week 204: number analyzed (Participants) | 53
  Week 204 | 34
  Week 216: number analyzed (Participants) | 53
  Week 216 | 32
  Week 228: number analyzed (Participants) | 45
  Week 228 | 20
  Week 240: number analyzed (Participants) | 29
  Week 240 | 13
  Week 252: number analyzed (Participants) | 23
  Week 252 | 10

3. Primary Outcome: Part 1: Number of Participants With Improvement in Simple Endoscopic Score for Crohn's Disease (SES-CD) Score at Week 108
Description: SES-CD is an endoscopic score composite of 4 variables (ulcers size, percentage of ulcerated surface, inflamed surface, and presence of narrowing) in up to 5 ileocolonic segments (ileum right, colon, transverse colon, left colon, rectum) and scored on a scale of 0-3, with total score from 0-60. Higher score indicates higher ulcer surface/size in the 4 variables. Endoscopic improvement was defined as ≥50% reduction in SES-CD score compared to baseline.
Time Frame: At OLE Week 108
Population: OLE population included all participants who received at least one dose of study drug in Study GA29145 Part 1 (OLE). Overall number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 242
Participants | 147

4. Primary Outcome: Part 1: Number of Participants With Adverse Event (AE) and Severity of AEs as Assessed Using National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. AEs were graded as per NCI CTCAE v4.0. Grade 1=Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3=Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4=Life threatening consequences, urgent intervention indicated; Grade 5=Death related to AE. Multiple occurrences of AEs in the same category at the worst (highest) NCIC-CTCAE grade for an individual are counted only once.
Time Frame: From Day 1 up to end of 12-week safety follow-up in OLE (approximately 6.3 years)
Population: OLE population included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants
  AEs, Any Grade | 624
  Grade 1 AEs | 121
  Grade 2 AEs | 259
  Grade 3 AEs | 214
  Grade 4 AEs | 27
  Grade 5 AEs | 3

5. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigation, whether or not considered related to the medicinal (investigational) product. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years)
Population: OLE popuation included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants | 206

6. Primary Outcome: Part 1: Number of Participants With Infection Related AEs and Severity of Infection-Related AEs Assessed Using NCI CTCAE v4.0
Description: AE=untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. AEs were graded per NCI CTCAE v4.0. Grade 1=Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3=Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living; Grade 4=Life-threatening consequences/urgent intervention indicated; Grade 5=Death related to adverse event. If a participant experienced multiple occurrences of AEs at different grades, they were counted in each grade where they had at least one AE of that grade.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years)
Population: OLE population included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants
  Infection Related AEs, Any Grade | 366
  Grade 1 Infection Related AEs | 239
  Grade 2 Infection Related AEs | 194
  Grade 3 Infection Related AEs | 56
  Grade 4 Infection Related AEs | 5
  Grade 5 Infection Related AEs | 1

7. Primary Outcome: Part 1: Incidence Rate of Infection-related Adverse Event
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. AE rate (per 100 participant years) = [Total number of AEs (in OLE only) / Total number of participant years at risk (in OLE only)]*100. Total participant-years at risk is the sum over all participants of the time intervals (in years) from the first dose of study treatment in Part 1 (OLE) until the participant completes/withdraws from the study (including the 12-week safety follow-up, if applicable).
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years)
Population: OLE population included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Number (95% Confidence Interval); unit: event per 100 participant-years
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
event per 100 participant-years | 62.74 [58.74 to 66.94]

8. Primary Outcome: Part 1: Number of Participants With Serious Infection Related AES
Description: as for outcome 5
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years)
Population: OLE popuation included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants | 58

9. Primary Outcome: Part 1: Number of Participants With Injection Site Reactions and Severity of Injection Site Reactions Assessed Using NCI CTCAE v4.0
Description: AE=untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. Injection-site reaction=any local reaction occurring at the site of injection following study drug administration. Signs (e.g., erythema, induration/swelling at injection site) and symptoms (e.g., pain, pruritus at injection site). Injection site reactions were graded per NCI CTCAE v4.0. Grade 1=Tenderness with or without associated symptoms (e.g., warmth, erythema, itching); Grade 2=Pain; lipodystrophy; edema; phlebitis; Grade 3=Ulceration or necrosis; severe tissue damage; operative intervention indicated; Grade 4=life-threatening consequences or urgent intervention indicated; Grade=5 death related to AE.
Time Frame: From Day 1 up to end of safety 12-week follow-up in OLE (approximately 6.3 years)
Population: OLE population included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants
  Injection Site Reaction, Any Grade | 15
  Injection Site Reaction, Grade 1 | 14
  Injection Site Reaction, Grade 2 | 1
  Injection Site Reaction, Grade 3 | 0
  Injection Site Reaction, Grade 4 | 0
  Injection Site Reaction, Grade 5 | 0

10. Primary Outcome: Part 1: Number of Participants With Adverse Events Leading to Etrolizumab Discontinuation
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. Number of participants who discontinued etrolizumab treatment during the OLE period have been reported here.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years)
Population: OLE population included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants | 112

11. Primary Outcome: Part 1: Number of Participants With Malignancies
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. Number of participants who developed malignancies during the OLE period have been reported here.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years)
Population: OLE population included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants | 18

12. Primary Outcome: Part 1: Incidence Rate of Malignancies
Description: Malignancy rate (per 100 participant years) = [Total number of malignancies (in OLE only) / Total number of participant years at risk (in OLE only)]*100. Total participant-years at risk is the sum over all participants of the time intervals (in years) from the first dose of study treatment in Part 1 (OLE) until the participant completes/withdraws from the study (including the 12-week safety follow-up, if applicable).
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years)
Population: OLE population included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Number (95% Confidence Interval); unit: events per 100-participant-years
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
events per 100-participant-years | 1.85 [1.22 to 2.70]

13. Primary Outcome: Part 1: Number of Participants With Hypersensitivity Reactions and Severity of Hypersensitivity Assessed Using NCI-CTCAE v4.0
Description: Hypersensitivity was reported using the MedDRA anaphylactic reaction standard MedDRA query (SMQ) and Sampson's criteria. Hypersensitivity was assessed as per NCI CTCAE v4.0. Grade 1 = Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated; Grade 2 = Moderate; minimal, local or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3 = Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years)
Population: OLE population included all participants who received at least one dose of study drug in study GA29145 Part 1 (OLE).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 751
Participants
  Hypersensitivity Reactions, Any Grade | 3
  Hypersensitivity Reactions, Grade 1 | 2
  Hypersensitivity Reactions, Grade 2 | 0
  Hypersensitivity Reactions, Grade 3 | 1

14. Primary Outcome: Part 2: Number of Participants With Confirmed or Suspected Progressive Multifocal Leukoencephalopathy (PML)
Description: PML was assessed by the PML Subjective Checklist (symptom assessment) and the PML Objective Checklist (neurologic evaluation).
Time Frame: From end of safety follow-up in Part 1 or study GA29144 up to maximum of 92 weeks
Population: PML SM population included all participants who entered the PML SM phase. No treatment was administered in PML SM period, and hence participants entering from Part 1 (OLE) and the parent study have been reported together.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: PML-SM: Participants from Part 1 (OLE) and from the study GA29144 who were not eligible/did not wish to enroll in Part 1 (OLE) and had completed the 12-week safety follow-up period were enrolled in Part 2 (PML SM). Participants were monitored for PML for a maximum of 92-weeks, during which no etrolizumab treatment was administered.
Arm/Group | Part 2: PML-SM
Number analyzed (Participants) | 359
Participants | 0

ADVERSE EVENTS:
Time Frame: Part 1 (OLE): From Day 1 up to end of 12-week safety follow up in OLE (approximately 6.3 years); Part 2 (PML SM): From end of safety follow-up in Part 1 or in study GA29144 up to a maximum of 92-weeks
Description: OLE population included all participants who received at least one dose of open label etrolizumab in Part 1 of the study. PML SM population included all participants who entered the PML SM period. Part 2: PML SM arm includes all participants who entered Part 2 (PML SM) from Part 1 (OLE) or from the parent study GA29144. No treatment was administered in PML SM period, and hence participants entering from Part 1 (OLE) and the parent study have been reported together.
Groups:
- Part 2 (PML SM): Participants from Part 1 (OLE) and from the study GA29144 who were not eligible/did not wish to enroll in Part 1 (OLE) and had completed the 12-week safety follow-up period were enrolled in Part 2 (PML SM). Participants were monitored for PML for a maximum of 92-weeks, during which no etrolizumab treatment was administered.
Arm/Group | Part 1 (OLE): Etrolizumab | Part 2 (PML SM)
All-Cause Mortality (participants affected / at risk) | 3/751 | 1/359
Serious Adverse Events (participants affected / at risk) | 206/751 | 1/359
Other Adverse Events (participants affected / at risk) | 453/751 | 2/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (OLE): Etrolizumab (N=751) | Part 2 (PML SM) (N=359)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual field defect (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 5 (10) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 69 (84) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 5 (6) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 10 (12) | 0 (0)
Small intestinal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Granulomatous liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 7 (7) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 13 (14) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Measles (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 3 (3) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Varicella meningitis (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lisfranc fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Pregnancy test negative (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (3) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Septal panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Ileostomy closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Intestinal resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Neurosurgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Parenteral nutrition (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (OLE): Etrolizumab (N=751) | Part 2 (PML SM) (N=359)
Anaemia (Blood and lymphatic system disorders) | 42 (52) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 82 (109) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 174 (229) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 53 (68) | 0 (0)
Nausea (Gastrointestinal disorders) | 52 (63) | 0 (0)
Vomiting (Gastrointestinal disorders) | 43 (52) | 0 (0)
COVID-19 (Infections and infestations) | 80 (81) | 0 (0)
Nasopharyngitis (Infections and infestations) | 80 (136) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 58 (80) | 0 (0)
Urinary tract infection (Infections and infestations) | 38 (46) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 87 (119) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 43 (52) | 0 (0)
Headache (Nervous system disorders) | 76 (96) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT02403323/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT02403323/SAP_001.pdf